CLINICAL TRIAL: NCT03789773
Title: Holographic Mm-wave Imaging in Radiation Oncology
Brief Title: Holographic Mm-Wave Imaging in Patients Undergoing Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant ended, no accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0S-18-6; NCI-2018-02994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-18-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-08

CONDITIONS: Unspecified Adult Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (holographic mm-wave imaging) (Experimental): Patients undergo holographic mm-wave imaging in radiotherapy treatment position after initial CT simulation.
  Interventions: Device: Millimeter-Wave Holographic Imaging

INTERVENTIONS:
Device: Millimeter-Wave Holographic Imaging — Undergo mm-wave holographic imaging
  Other Names: Holographic Millimeter-wave Imaging; Holographic mm-Wave Imaging; MMW Holographic Imaging; Millimeter-wave Imaging; MMW Imaging; MMW

SUMMARY:
This trial studies the quality of holographic mm-wave imaging in patients undergoing radiation therapy. Holographic mm-wave imaging is a common type of imaging used in airport body scanners that may be helpful in improving the efficiency and positioning of radiation oncology patients and their overall experience.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain patient images in a clinical setting and assess their quality.

SECONDARY OBJECTIVES:

I. To assess the registration agreement through a voxel-voxel distance-to-agreement metric.

OUTLINE:

Patients undergo holographic mm-wave imaging in radiotherapy treatment position after initial computed tomography (CT) simulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to receive either an optical or CBCT imaging scan as part of their treatment management.
* The study will be open to English and Spanish speaking participants.

Exclusion Criteria:

* Patients that are not scheduled for fluoroscopic or optical imaging as part of the normal course of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of holographic image quality | Up to 1 year
  Qualitative assessment of image quality by study physicians according to the scoring of each image as: 1 = High Quality (A); 2= Acceptable Quality (B); 3 = Poor/Unacceptable Quality (C). Lower value (1) represents a better score than higher value (3). There are no subscales and or total scores. The quality scores of the images will be tabulated.

SECONDARY OUTCOMES:
Image registration agreement between mm-wave holographic images and a cone-beam computed tomography (CBCT)/optical surface image | Up to 1 year
  The distribution of the percent of points in voxel-voxel analysis to agree to better than 2 mm will be tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reilly, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States